CLINICAL TRIAL: NCT01635413
Title: Group Exercise Training for Functional Improvement After Treatment (The GET FIT Trial)
Acronym: GET FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kerri Winters, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00008560; NCI-2012-01141 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MR00045870; CPC-12080-LX; IRB00008560 (Other: OHSU Knight Cancer Institute); R01CA163474 (NIH)
Record Dates: First submitted 2012-06-29; First posted 2012-07-09 (Estimated); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Malignant Neoplasm; Postmenopausal
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (strength training) (Experimental): Patients attend strength training classes for 1 hour 2 days per week.
  Interventions: Behavioral: Exercise Intervention; Other: Questionnaire Administration
- Arm II (tai chi) (Experimental): Patients attend tai chi classes for 1 hour 2 days per week.
  Interventions: Behavioral: Exercise Intervention; Other: Questionnaire Administration
- Arm III (control) (Active Comparator): Patients attend supervised stretching and relaxation classes for 1 hour 2 days per week.
  Interventions: Behavioral: Exercise Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Exercise Intervention — Undergo strength training classes
  Arms: Arm I (strength training)
Behavioral: Exercise Intervention — Undergo tai chi classes
  Arms: Arm II (tai chi)
Behavioral: Exercise Intervention — Undergo stretching and relaxation classes
  Arms: Arm III (control)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research is being done to compare the physical and quality of life benefits of two different types of exercise- tai chi versus strength training- for female cancer survivors who have had chemotherapy. Each exercise- tai chi and strength training- will be compared to participants in a group that performs flexibility and relaxation exercises, which is expected to have different benefits than either tai chi or strength training.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the relative efficacy of tai chi and strength training to prevent falls in female cancer survivors.

II. Determine the mechanism by which tai chi and strength training each reduces the risk of falls.

III. Determine how well the benefits of each intervention persist after structured training stops.

SECONDARY OBJECTIVE:

I. Evaluate the effect of the intervention on physical functioning.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients attend strength training classes for 1 hour 2 days per week.

ARM II: Patients attend tai chi classes for 1 hour 2 days per week.

ARM III: Patients attend supervised stretching and relaxation classes for 1 hour 2 days per week.

In all arms, treatment continues for 6 months.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage I-III cancer other than cancers of the brain or spinal cord (confirmed by patient self-report on the Health History Questionnaire; if patient is unable to confirm either the site of her cancer or that her stage of cancer is < stage IV, we will send a letter to her physician to confirm this criterion)
* Completed chemotherapy > 3 months prior to enrollment and no concurrent adjuvant therapy other than hormone manipulation therapy for breast cancer (confirmed by patient self-report on the Health History Questionnaire; if patient is unable to confirm whether or not she completed chemotherapy 3 months prior to enrollment, we will send a letter to her physician to confirm eligibility on this criterion)
* Postmenopausal (confirmed by self-report on the Health History Questionnaire; menopausal status could also be confirmed by a recent [< 6 months from enrollment] laboratory report documenting serum follicle-stimulating hormone [FSH] > 30 mIU/ml and/or serum estradiol < 30 pg/ml)
* Currently underactive (< 60 minutes of moderate intensity exercise per week in the last month) (confirmed by self-report on the Health History Questionnaire)

Exclusion Criteria:

* Cognitive difficulties that preclude answering the survey questions, participating in the exercise classes or performance tests, or providing informed consent (confirmed by the professional opinion of the Principal Investigator, Dr. Kerri Winters-Stone)
* A medical condition, movement or neurological disorder, or medication use that contraindicates participation in moderate intensity exercise (confirmed by self-report on the Health History Questionnaire, and by physician clearance; if in the professional opinion of the Principal Investigator, Dr. Kerri Winters-Stone, contraindications other than those identified by the patient or physician are present, she may consider the participant ineligible)

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2012-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Falls | Baseline up to 12 months
  Prospective assessment of falls will be done by collecting monthly and quarterly reports returned by postal and/or electronic mail. A fall is defined as unintentionally coming to rest on the ground or at some other lower level, not as a result of a major intrinsic event (e.g., stroke or syncope) or overwhelming hazard.

SECONDARY OUTCOMES:
Muscle strength | Baseline, 3 and 6 months during study treatment and 6 months after completion of study treatment
  Measured by 1-repetition maximum (1-RM) for leg press. The maximum amount of weight that can be lifted one time.
Postural stability | Baseline, 3 and 6 months during study treatment and 6 months after completion of study treatment
  Measured by Computerized dynamic posturography using the sensory organization test (SOT) and limits of stability (LOS). The SOT generates an equilibrium scores and sensory ratios that range from 0-100, where 100 = perfect stability and 0 = an inability to maintain balance and a fall. The LOS measures the average % of targeted distances reached (end point excursion) and average % of movement in the targeted direction (directional control).
Flexibility | Baseline, 3 and 6 months during study treatment and 6 months after completion of study
  Measured by the standardized chair sit-and-reach test for lower body flexibility. Designed for older adults with demonstrated validity and reliability in older adults (test-retest 0.95-0.96).
Physical Function | Baseline, 3 and 6 months during study treatment and 6 months after completion of study
  Measured by the Physical Performance Battery (PPB). The PPB consists of 3 timed tests: 5 repeated chair stands, standing balance, and gait speed over 4 meters. Each test is scored 0 (unable) to 4 (completes without difficulty), based on quartiles of performance, then scores are summed. The possible range of scores is 0-12.
Injurious falls | Baseline up to 12 months
  Collected during prospective monthly and quarterly reports of falls. A fall is considered ''injurious'' if it results in fractures, head injuries, sprains, bruises, scrapes, or serious joint injuries, or if the participant seeks medical care.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Winters-Stone, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Derived] Sitemba J, Crisafio M, Li F, Eckstrom E, Winters-Stone KM. Evaluating recruitment, retention, and adherence patterns in the GET FIT fall prevention exercise trial in older, postmenopausal cancer survivors. Support Care Cancer. 2025 Jul 28;33(8):727. doi: 10.1007/s00520-025-09767-1. PMID 40721864
- [Derived] Winters-Stone KM, Stoyles SA, Dieckmann NF, Eckstrom E, Luoh SW, Horak FB, Roeland EJ, Li F. Can strength training or tai ji quan training reduce frailty in postmenopausal women treated with chemotherapy? A secondary data analysis of the GET FIT trial. J Cancer Surviv. 2024 Aug;18(4):1179-1189. doi: 10.1007/s11764-024-01592-5. Epub 2024 Apr 20. PMID 38642204
- [Derived] Winters-Stone KM, Roeland EJ, Li F, Eckstrom E, Horak F, Dieckmann NF, Stoyles SA, Luoh SW. Reply to Y.-T. Hu et al. J Clin Oncol. 2023 Sep 10;41(26):4316-4317. doi: 10.1200/JCO.23.01034. Epub 2023 Jun 28. No abstract available. PMID 37379504
- [Derived] Winters-Stone KM, Horak F, Dieckmann NF, Luoh SW, Eckstrom E, Stoyles SA, Roeland EJ, Li F. GET FIT: A Randomized Clinical Trial of Tai Ji Quan Versus Strength Training for Fall Prevention After Chemotherapy in Older, Postmenopausal Women Cancer Survivors. J Clin Oncol. 2023 Jun 20;41(18):3384-3396. doi: 10.1200/JCO.22.01519. Epub 2023 Mar 8. PMID 36888933
- [Derived] McGinnis GJ, Holden S, Yu B, Ransom C, Guidarelli C, De B, Diao K, Boyce D, Thomas CR Jr, Winters-Stone K, Raber J. Association of fall rate and functional status by APOE genotype in cancer survivors after exercise intervention. Oncotarget. 2022 Nov 17;13:1259-1270. doi: 10.18632/oncotarget.28310. PMID 36441715
- [Derived] Winters-Stone KM, Li F, Horak F, Luoh SW, Bennett JA, Nail L, Dieckmann N. Comparison of tai chi vs. strength training for fall prevention among female cancer survivors: study protocol for the GET FIT trial. BMC Cancer. 2012 Dec 5;12:577. doi: 10.1186/1471-2407-12-577. PMID 23217054